CLINICAL TRIAL: NCT06193291
Title: Effect of Hot Water Immersion on Heart Rate Variability (HRV) and Glucose
Brief Title: Effect of Hot Water Immersion on Heart Rate Variability and Glucose
Acronym: HWI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Principal Investigator, Jeff Moore, Principal Investigator, San Diego State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Hot Water Immersion
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Glucose Tolerance; HRV

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Thermoneutral (No Intervention): Participant sits at room temperature during an oral glucose tolerance test
- Feet heating (Experimental): Participant sits with feet placed in hot water during an oral glucose tolerance test
  Interventions: Procedure: Feet heating
- Calf heating (Experimental): Participant sits with legs, up to calves, placed in hot water during an oral glucose tolerance test
  Interventions: Procedure: Calf heating

INTERVENTIONS:
Procedure: Feet heating — Feet placed in hot water
  Arms: Feet heating
Procedure: Calf heating — Feet to calves placed in hot water
  Arms: Calf heating

SUMMARY:
Heat therapy has been shown to reduce risk of various diseases, including heart disease, alzheimers, and pneumonia, as well as all-cause mortality . A previous study found heating a single hand lowers postprandial blood glucose levels with a magnitude similar to certain exercise interventions such as 40 minutes of slow walking We propose that heating both feet and heating both legs up to the calves will result in similar glucose reductions in a dose response manner.Overview To determine the effect of heating both feet to the ankles and heating both legs to the calves on postprandial blood glucose

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years

Exclusion Criteria:

* previously diagnosed diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Blood Glucose | 120 min

SECONDARY OUTCOMES:
Heart rate variability | 120 min

CONTACTS AND LOCATIONS:
Locations (1):
- San Diego State University, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Laukkanen JA, Laukkanen T, Kunutsor SK. Cardiovascular and Other Health Benefits of Sauna Bathing: A Review of the Evidence. Mayo Clin Proc. 2018 Aug;93(8):1111-1121. doi: 10.1016/j.mayocp.2018.04.008. PMID 30077204
- [Background] Kimball AL, McCue PM, Petrie MA, Shields RK. Whole body heat exposure modulates acute glucose metabolism. Int J Hyperthermia. 2018;35(1):644-651. doi: 10.1080/02656736.2018.1516303. Epub 2018 Oct 10. PMID 30303421
- [Background] Moore J, Kressler J, Buono MJ. Hand heating lowers postprandial blood glucose concentrations: A double-blind randomized controlled crossover trial. Complement Ther Med. 2020 Mar;49:102280. doi: 10.1016/j.ctim.2019.102280. Epub 2019 Dec 12. PMID 32147036